CLINICAL TRIAL: NCT04304053
Title: Treatment of Non-severe Confirmed Cases of COVID-19 and Chemoprophylaxis of Their Contacts as Prevention Strategy: a Cluster Randomized Clinical Trial (PEP CoV-2 Study)
Brief Title: Treatment of COVID-19 Cases and Chemoprophylaxis of Contacts as Prevention
Acronym: HCQ4COV19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Department of Health, Generalitat de Catalunya (Other Government); Laboratorios Gebro Pharma SA (Unknown); Laboratorios Rubió (Unknown); Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Oriol Mitja, Prof (Ass) Infectious Disease and Global Health, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCQ4COV19; 2020-001031-27 (EudraCT Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Primary study: Cluster-randomized clinical trial of Covid-19 contacts
  Secondary study: Randomized clinical trial of Covid-19 cases
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention- SARS-CoV-2 surveillance (Active Comparator): Study 1- Contacts will complete a survey collecting demographic, epidemiological and clinical data and provides a swab for RT-PCR testing at baseline and day 14.
  Study 2- Index case completes a survey collecting demographic, epidemiological and clinical data and provides a swab for RT-PCR testing at baseline and on days 3 and 7.
  Isolation of patient and contact tracing as per national guidelines.
  Interventions: Other: Standard Public Health measures
- Testing, treatment and prophylaxis of SARS-CoV-2 (Experimental): Study 1- Contacts receive Hydroxychloroquine prophylaxis. Contacts will complete a survey collecting demographic, epidemiological and clinical and provides a swab for RT-PCR testing at baseline and day 14.
  Study 2- Index case receives Hydroxychloroquine. Index case completes a survey collecting demographic, epidemiological and clinical data and provides a swab for RT-PCR testing at baseline and on days 3, and 7.
  Isolation of patient and contact tracing as per national guidelines.
  Interventions: Drug: Treatment and prophylaxis; Other: Standard Public Health measures

INTERVENTIONS:
Drug: Treatment and prophylaxis — Cases will be offered a therapeutic regimen hydroxychloroquine (200mg tablets) 800mg on day 1, and 400mg on days 2-7
  Contacts will be offered a prophylactic regimen of hydroxychloroquine (200mg tablets) 800mg on day 1, and 400mg on days 2-7.
  Arms: Testing, treatment and prophylaxis of SARS-CoV-2
Other: Standard Public Health measures — Isolation of patient and contact tracing as per national guidelines.

SUMMARY:
This study is a research project to evaluate the efficacy of hydroxychloroquine for post-exposure prophylaxis and early treatment of Covid-19. The intervention entails administering prophylactic hydroxychloroquine to all contacts (Study 1) and treating non severe confirmed cases with hydroxychloroquine (Study 2).

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ) is a drug that has been extensively used for the prevention of malaria. HCQ showed excellent in vitro results and strong antiviral effects on SARS-CoV-2 infection of primate cells at low concentration. Empirical data for the efficacy of HCQ in hospitalized Covid-19 patients became available after the start of this study; HCQ administration did not result in a significantly higher PCR negative conversion in a RCT including 150 patients and there was no reduction in the risk of death/intubation in two large observational studies.

Study 1 -We investigated the efficacy and safety of HCQ to prevent secondary SARS-CoV-2 infection and Covid-19 disease in contacts exposed to a PCR-positive Covid-19 case during.

Study 2- We also conducted a study to test the hypothesis that HCQ treatment would be more efficacious than no-treatment for patients with mild Covid-19.

Initially, the protocol included the use of combined treatment with a HIV protease inhibidor (cobicistat-boosted darunavir) for cases (study 2), but it was adapted to HCQ alone after the recommendation of the pharmaceutical company not to use DRVc for the treatment of Covid-19 due to lack of activity in-vitro.

ELIGIBILITY:
Study 1:

Inclusion Criteria for a contact:

1. Asymptomatic individuals exposed to a PCR confirmed COVID19 case within 7 days as either a healthcare worker or household contact
2. Aged ≥18 years male or female;
3. In women of childbearing potential, negative pregnancy test and commitment to use contraceptive method throughout the study.
4. Willing to take study medication;
5. Willing to comply with all study procedures;
6. Able to provide oral, informed consent and/or assent.

Exclusion Criteria for a contact:

1. With known history of cardiac arrhythmia (or QT prolongation syndrome);
2. Unable to take drugs by mouth;
3. With significantly abnormal liver function (Child Pugh C)
4. Need of dialysis treatment, or GFR≤30 mL/min/1.73 m2;
5. Participants with psoriasis, myasthenia, haematopoietic and retinal diseases,CNS-related hearing loss or glucose-6-phosphate dehydrogenase deficit;
6. Persons already treated with any of the study drugs during the last 30 days;
7. Pregnant or lactating women;
8. Any contraindications as per the Data Sheet of Hydroxychloroquine.

Study 2:

Inclusion Criteria for a case:

1. Patients who meet the requirements of the New Coronavirus Infection Diagnosis (Acute <5 days respiratory infection symptoms, or fever alone, or acute cough alone and positive PCR)
2. Aged ≥18 years male or female;
3. In women of childbearing potential, negative pregnancy test and commitment to use contraceptive method throughout the study.
4. Willing to take study medication
5. Willing to comply with all study procedures, including repeat nasal swab at day 3
6. Able to provide oral and written informed consent

Exclusion Criteria for a case:

1. Hospital admission
2. Serious condition meeting one of the following: (1) respiratory distress with respiratory rate >=30 breaths/min; (2) oxygen saturation<=93% on quiet status; (3) Arterial partial pressure of oxygen (PaO2)/oxygen concentration<=300mmHg;
3. Critically ill patients meeting one of the following: (1) Experience respiratory failure and need to receive mechanical ventilation; (2) Experience shock; (3) Complicated with other organs failure and need intensive care and therapy in ICU;
4. Participants under treatment with medications likely to interfere with experimental drugs
5. Unable to take drugs by mouth;
6. With significantly abnormal liver function (Child Pugh C)
7. Need of dialysis treatment, or GFR≤30 mL/min/1.73 m2;
8. Participants with psoriasis, myasthenia, haematopoietic and retinal diseases,CNS-related hearing loss or glucose-6-phosphate dehydrogenase deficit
9. Participants with severe neurological and mental illness;
10. Pregnant or lactating women;
11. Inability to consent and/or comply with study protocol;
12. Individuals with known hypersensitivity to the study drugs.
13. Persons already treated with any of the study drugs during the last 30 days.
14. Any contraindications as per the Data Sheet of Hydroxychloroquine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Study 1- Clinical and virological outcome in exposed contacts | Up to 14 days after start of treatment
  Incidence of secondary PCR confirmed symptomatic Covid-19 episodes among contacts after high risk PCR+ exposure
Study 1- Transmission of SARS-CoV-2 in exposed contacts | Up to 14 days after start of treatment
  Incidence of symptomatically compatible or a PCR-positive result regardless of symptoms
Study 2- Virological outcome in index cases | Up to 7 days after start of treatment
  Reduction of viral RNA load in nasopharyngeal swabs at days 3, and 7 after treatment start.
Study 2- Clinical outcome in index cases | Up to 28 days after start of treatment
  Time from randomization to complete resolution of symptoms at an extended 28-days follow-

CONTACTS AND LOCATIONS:
Locations (1):
- Departament de Salut, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Open access
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 30 days after start of treatment
Access Criteria: Open access for everybody
URL: http://www.estudicovid19.org

REFERENCES:
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583
- [Derived] Mitja O, Corbacho-Monne M, Ubals M, Alemany A, Suner C, Tebe C, Tobias A, Penafiel J, Ballana E, Perez CA, Admella P, Riera-Marti N, Laporte P, Mitja J, Clua M, Bertran L, Sarquella M, Gavilan S, Ara J, Argimon JM, Cuatrecasas G, Canadas P, Elizalde-Torrent A, Fabregat R, Farre M, Forcada A, Flores-Mateo G, Lopez C, Muntada E, Nadal N, Narejos S, Nieto A, Prat N, Puig J, Quinones C, Ramirez-Viaplana F, Reyes-Uruena J, Riveira-Munoz E, Ruiz L, Sanz S, Sentis A, Sierra A, Velasco C, Vivanco-Hidalgo RM, Zamora J, Casabona J, Vall-Mayans M, Gonzalez-Beiras C, Clotet B; BCN-PEP-CoV2 Research Group. A Cluster-Randomized Trial of Hydroxychloroquine for Prevention of Covid-19. N Engl J Med. 2021 Feb 4;384(5):417-427. doi: 10.1056/NEJMoa2021801. Epub 2020 Nov 24. PMID 33289973